CLINICAL TRIAL: NCT06312553
Title: Remotely Delivered Mindfulness-Based Diabetes Education for Rural Adults With Uncontrolled Diabetes and Elevated Distress
Brief Title: Remotely Delivered Mindfulness-Based Diabetes Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Caroline Presley, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-300012515; P50MD017338 (NIH)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Distress; Glycemic Control; Remote Patient Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Remotely delivered Mindfulness-Based Diabetes Education with remote patient monitoring (Experimental): The Mindfulness-Based Diabetes Education (MBDE) program will be delivered in 8, 2-hour weekly sessions, then 2 booster sessions, total duration of 6 months. MBDE will be delivered over Zoom with content delivered by the interventionist per the program manual. Participants will be provided with a tablet and WIFI hotspot. Sessions will be video-recorded and made available to participants in case of missed sessions.
  Interventions: Behavioral: Remotely delivered Mindfulness-Based Diabetes Education with remote patient monitoring
- Standard Diabetes Self Management Education (Active Comparator): Standard DSME will be delivered by a certified diabetes educator in four biweekly sessions of 2 hours duration; topics will include healthy eating, physical activity, medication usage, self-monitoring, preventing and managing complications, healthy coping, and problem solving.18 Standard DSME will be delivered in groups of 8-12 participants via Zoom.
  Interventions: Behavioral: Standard Diabetes Self Management Education

INTERVENTIONS:
Behavioral: Remotely delivered Mindfulness-Based Diabetes Education with remote patient monitoring — Remotely delivered Mindfulness-Based Diabetes Education with remote patient monitoring described in study arm
  Arms: Experimental: Remotely delivered Mindfulness-Based Diabetes Education with remote patient monitoring
Behavioral: Standard Diabetes Self Management Education — Standard Diabetes Self Management Education described in study arm
  Arms: Standard Diabetes Self Management Education

SUMMARY:
Diabetes distress is common affecting over one-third of people with type 2 diabetes, negatively impacting self-management and outcomes, and disproportionately affecting low-income individuals. The proposed project will conduct a pilot randomized controlled trial comparing remotely delivered Mindfulness-Based Diabetes Education plus remote patient monitoring of blood glucose to standard Diabetes Self-Management Education in rural Black adults with type 2 diabetes and elevated diabetes distress who receive care within federally qualified health centers to assess feasibility and acceptability.

DETAILED DESCRIPTION:
For Aim 2, investigators will conduct a pilot randomized controlled trial (RCT) comparing Mindfulness-Based Diabetes Education to standard Diabetes Self-Management Education in rural, Black adults with uncontrolled type 2 diabetes and elevated diabetes distress. Pilot RCT participants will be recruited from Federally Qualified Health Centers in the rural Black Belt region of Alabama. Participants will be recruited through opt-out letters and phone calls to adults with diabetes seen within the preceding two years at study sites, as well as through in-person recruitment during clinic or through direct referral by provider or patient.

Investigators plan to recruit up to 80 participants total, 40 per study arm. Investigators will obtain screening consent prior to conducting screening diabetes distress and A1C (per previously described inclusion criteria). Informed consent will be obtained from eligible participants prior to enrollment or randomization. Participants will be randomly assigned to receive either Mindfulness-Based Diabetes Education or standard Diabetes Self-Management Education on a 1:1 basis; randomization will be stratified by study site and sex.

The Mindfulness-Based Diabetes Education intervention will be delivered remotely by Zoom videoconference in 8 weekly sessions in a group setting. Following completion of the 8-week program, participants will receive 2 bimonthly individual booster sessions by phone for a total duration of 6 months. Mindfulness-Based Diabetes Education will be delivered by an interventionist, who is a nurse practitioner with clinical expertise in diabetes care and education as well as training in MBSR. During intervention sessions, participants will be introduced to different mindfulness practices, including awareness of breath meditation, body scan exercise, walking meditation, and mindful yoga, and informal practices including the application of mindfulness to daily activities. Additionally, participants will receive instruction and have opportunities to practice bringing mindful attention to specific diabetes self-management behaviors. For example, a session will include exploration of mind-body connections, instruction of walking meditation, educational module on physical activity (PA), and a PA exercise with mindful attention. Participants will be asked to complete daily home mindfulness exercises and self-monitoring of diabetes self-management behaviors. Mindfulness-Based Diabetes Education will use incremental goal setting with self-monitoring, feedback, and modeling to build participants' self-efficacy and on development of social support. Sessions will include time for participants to set SMART goals. Additionally, participants in the intervention arm will receive a glucometer and kit to facilitate remote monitoring of blood glucose. Participants will be instructed to measure blood glucose levels at least 1 time per day.

Standard DSME will be delivered by a Certified Diabetes Educator remotely by Zoom videoconference in 4 biweekly, 2-hour sessions. DSME sessions will cover seven core content areas including healthy eating, physical activity, medication usage, self-monitoring, preventing and treating acute and chronic complications, healthy coping, and problem solving.

The primary outcomes of the study will be acceptability and feasibility. Participants in the Mindfulness-Based Diabetes Education arm will be asked to participate in a semi-structured interview to assess the acceptability of the intervention including participants' perspectives on intervention content; perceived benefits or negative effects of the intervention; appropriateness of intervention duration and frequency; satisfaction with interventionist; satisfaction with intervention content; barriers to engagement; suggestions to improve the intervention; and overall satisfaction. Feasibility of delivering Mindfulness-Based Diabetes Education will be assessed through process measures including: percentage of screened participants who are eligible; percentage of eligible participants who enroll; ability to randomize participants to study arms; representativeness of participants by age, gender, and race/ethnicity; number of sessions attended; participant adherence to study tasks, including home mindfulness exercises and self-monitoring of diabetes self-management behaviors; barriers to participation in intervention sessions or completing study activities at home; reasons for dropping out; and overall study retention. This study will also provide an opportunity to test the feasibility of recruitment strategies, allocation procedures, and assessment procedures and measures.

Participants will complete assessments at baseline and 6 months, which will include an interviewer-administered questionnaire of participant characteristics and validated measures of stress and diabetes distress, mood, diabetes self-management behaviors, self-efficacy, social needs, and health related-quality of life Participants will have height and weight measured, as well as point-of-care hemoglobin A1c (A1C) testing at baseline and 6 months. Outcome assessors will be blinded to the study arm to which participants are assigned.

ELIGIBILITY:
Inclusion Criteria:

* age 19 years or older
* diagnosis of type 2 diabetes
* Black race (self-report)
* receipt of care at one of the study sites with one or more visits to within the prior year
* presence of elevated diabetes distress (score ≥2 on Diabetes Distress Scale indicating moderate-severe distress)
* uncontrolled diabetes indicated by an elevated hemoglobin A1c (A1C) ≥8%

Exclusion Criteria (Presence of any of the following criteria):

* non-English speaker
* current pregnancy
* diagnosis of a severe psychiatric comorbidity including bipolar disorder, schizophrenia, or a history of psychosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: percentage of screened participants who are eligible | 6 months
  Investigators will assess the percentage of screened participants who are eligible to participate in the study. Study staff will track the number of participants who are screened for participation and the number of participants who are eligible to participate.
Feasibility: percentage of eligible participants who enroll | 6 months
  Investigators will assess the percentage of eligible participants who enroll in the study. Study staff will track the number of participants who are eligible for participation and the number of participants who enroll in the study.
Feasibility: ability to randomize participants to study arms | 6 months
  Investigators will assess the percentage of eligible participants who are randomized. Study staff will track the number of participants who are enrolled and the number of participants who are randomized.
Feasibility: distribution of participants by demographics | 6 months
  Investigators will collect demographics of study participants, including age and gender by participant self-report. This information will be obtained during a questionnaire administered to participants in English by a trained interviewer. Investigators will use descriptive statistics to characterize the demographics of the study sample.
Feasibility: percentage of sessions attended | 6 months
  Investigators will track the number of sessions attended by each participant and calculate the percentage of sessions attended by each participant.
Feasibility: participant adherence to study tasks include home mindfulness practices, self-monitoring activities. | 6 months
  At each session, Investigators will collect logs of participants' home mindfulness and self-monitoring activities. Investigators will calculate participant adherence to recommended activities for each participant.
Feasibility: barriers to participation in intervention sessions or completing study activities at home | 6 months
  Investigators will collect information from participants to assess any barriers they experienced attending study sessions or completing recommended home activities. This information will be obtained during a questionnaire administered to participants in English by a trained interviewer.
Feasibility: reasons for dropping out | 6 months
  Investigators will collect information from participants who drop out of the intervention or study regarding the reason for dropping out.
Feasibility: overall study retention | 6 months
  Investigators will track the number of participants who enroll in the study and complete assessments at each time point - baseline, 2 months, and 6 months.
Acceptability | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants. Including: perceived positive and negative effects, assessment of intervention content, appropriateness of duration and frequency, satisfaction with interventionist, barriers to engaging with intervention sessions or content, suggestions to improve the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Caroline A Presley, MD, MPH, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No